CLINICAL TRIAL: NCT03848689
Title: Fluoroquinolone Restriction Ofr the Prevention of C. Difficile Infection (CDI)_the FIRST Trial
Brief Title: FQ Restriction for the Prevention of CDI
Acronym: FIRST
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2018-0852; 1R01HS026226-01 (AHRQ); A534265 (Other: UW, Madison); SMPH/MEDICINE/MEDICINE*I (Other: UW, Madison); Protocol ver 5.0 20 Dec 2020 (Other: UW Madison)
Record Dates: First submitted 2018-10-02; First posted 2019-02-21 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Clostridium Difficile; Clostridium Difficile Infection; C Difficile Colitis
MeSH Terms: conditions — Clostridium Infections; Enterocolitis, Pseudomembranous

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FQ PPA Group: Fluoroquinolone Preprescription Authorization from Infection Control consult, once, prior to prescribing fluoroquinolone
  Interventions: Other: fluoroquinolone preprescription authorization
- Control Group: No preprescription authorization needed from Infection control prior to prescribing fluoroquinolone
  Interventions: Other: Control

INTERVENTIONS:
Other: fluoroquinolone preprescription authorization — Requires authorization from Infection Control consult prior to prescribing fluoroquinolone
  Other Names: FQ PPA
  Groups: FQ PPA Group
Other: Control — Does not require authorization from Infection Control prior to prescribing fluoroquinolone
  Other Names: No FQ PPA
  Groups: Control Group

SUMMARY:
This study evaluates the effectiveness of a new intervention, fluoroquinolone (FQ) Preprescription Authorization (PPA) strategy, to reduce and prevent Clostridium difficile infection (CDI) in hospital intensive care units (ICUs). The investigators will model a successful FQ PPA strategy in several Wisconsin ICUs and compare whether the intervention has improved outcomes in reducing CDIs. An additional goal of the study is to evaluate environmental and work system factors using systems engineering models in order to determine the most successful way to implement these new strategies.

DETAILED DESCRIPTION:
The objective of the proposed study is to evaluate the effectiveness and implementation of a fluoroquinolone (FQ) Preprescription Authorization (PPA) as an antibiotic stewardship (AS) strategy to target and prevent CDI, promote appropriate antibiotic use, and reduce the transmission of resistant bacteria. This will contribute to the long-term goal of reducing the burden of Clostridium difficile infection (CDI), which is an essential step in improving the safety and quality of healthcare. FQ PPA is a particularly promising AS strategy to reduce CDI. Although FQs are one of the most frequently utilized classes of antibiotics in inpatient acute care facilities and are closely associated with risk for CDI, FQ usage has not been the focus of control efforts in endemic settings in the US. The proposed study will use an effectiveness-implementation hybrid type 2 design to simultaneously evaluate the efficacy of an FQ PPA intervention to reduce CDI as well as the key considerations for implementing such an intervention successfully. Intensive care units in acute care hospitals throughout Wisconsin will participate in this stepped wedge cluster randomized controlled trial. The specific aims for the proposed study are to: 1) determine the impact of a FQ PPA on hospital-onset and healthcare-associated CDI rates and other clinical outcomes compared with usual care; and 2) evaluate the implementation of FQ PPA using a systems engineering approach. For aim 1, electronic health record data will be used to evaluate the impact of the FQ PPA on hospital-onset and healthcare-associated CDI, as well as other important clinical outcomes. For aim 2, surveys and interviews with healthcare providers will be used to evaluate the contextual, implementation, and work system factors that contribute to successful implementation of a FQ PPA intervention. In addition to addressing an urgent need to identify effective AS strategies, this study will provide a framework to implement and evaluate other interventions for healthcare-acquired infection (HAI) prevention. Regardless of the results, the proposed study will generate data, tools and methods with widespread applicability for AS initiatives in healthcare-associated infection prevention.

ELIGIBILITY:
Inclusion Criteria:

* Medical-surgical intensive care unit with at least 10 beds
* Presence of existing antibiotic stewardship (AS) program with pharmacist and ID physician support
* Electronic health record (EHR) vendor is Epic Systems Corporation
* Has ability to extract antibiotic usage data (days of therapy)
* Has ability to extract required outcomes data (CDI, mortality, length of ICU stay)
* Ability to extract or abstract data on indications for antibiotic use
* Adherence to best practices for infection control relevant to CDI

Exclusion Criteria:

* Medical-surgical intensive care units with a FQ restriction in place as part of their usual care procedures will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is comprised of clinicians and patients at 12 ICUs in 5 acute care hospitals. Once initiated, the intervention will be applied to all patients admitted to the ICU and all healthcare workers involved in antibiotic prescribing in that ICU.
Sampling Method: Probability Sample
Enrollment: 5871 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in the incidence of healthcare facility-onset Clostridiodes difficile infection (HO-CDI) with intensive care unit (ICU)-onset before and after initiating FQ PPA intervention | 24 Months
  Effectiveness of fluoroquinolone (FQ) Pre-prescription Authorization (PPA) intervention to reduce HO-CDI with ICU-onset will be assessed by comparing changes in incidence over pre- and post-intervention periods.
Change in the overall incidence of HO-CDI before and after initiating FQ PPA intervention | 24 months
  Effectiveness of FQ PPA intervention to reduce HO-CDI will be assessed by calculating changes in incidence over pre- and post-FQ PPA intervention periods.
Change in incidence of healthcare-associated CDI (HA-CDI) before and after initiation of FQ PPA intervention | 24 Months
  Effectiveness of FQ PPA intervention to reduce HA-CDI will be assessed by calculating changes in incidence over pre- and post-FQ PPA intervention periods.

SECONDARY OUTCOMES:
Change in the usage of FQ from the time of participant hospital admission per 1000 patient-days. | 24 months
  To confirm fidelity of implementation of FQ PPA intervention, the change in the usage of FQ and other antibiotics in days of therapy per 1000 patient-days will be measured.
Change in usage of non-FQ antibiotics per patient admission, and days of therapy per 1000 PD | 24 months
  To confirm fidelity of implementation of FQ PPA intervention, the change in the usage of antibiotics other than FQ in days of therapy per 1000 patient-days will be measured.
Change in the number of patients per site showing Acute Kidney Injury (AKI) using the Kidney Disease Improving Global Outcomes (KDIGO) guideline definition. | 24 months
  The potential of this intervention to increase usage of alternative antibiotics with a negative clinical outcomes such as AKI, as compared with usual care, will be measured by assessing change in incidence of AKI, defined as: Increase in serum creatinine by ≥ 0.3 mg/dl within 48 hours, or increase in serum creatinine to ≤1.5 times baseline or urine volume <0.5 mg/kg/hour for 6 hours.
Hospital Mortality Rate of Participants | 24 months
  Hospital mortality
Length of Participants's Hospital Stay | 24 months
  The impact of FQ PPA on negative clinical outcomes as compared with usual care by the length of hospital stay
Number of Participants Readmitted within 30 Days | 24 months
  The impact of FQ PPA intervention compared with usual care as it impacts the number of patients readmitted within 30 days.
Number of Incidences of Hospital Acquired Infections | 24 months
  The impact of FQ PPA on negative clinical outcomes as compared with usual care by the incidence of other, non-CDI hospital acquired infections.
Baseline proportion of CDI due to NAP-1 in site ICUs and associated facilities. | 24 months
  This would reflect whether the FQ PPA intervention was impacted by the prevalence of the strain of CDI most susceptible to FQ antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Nasia Safdar, MD PhD, Principal Investigator — University of Wisconsin, Madison
Locations (7):
- United States (7):
  - Mayo-Arizona, Phoenix, Arizona
  - Riverside University Health System Medical Center, Moreno Valley, California
  - Mayo-Rochester, Rochester, Minnesota
  - St. Luke's Health System, Kansas City, Missouri
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Gundersen Health Systems, La Crosse, Wisconsin
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Safdar N, Parmasad V, Brown R, Carayon P, Lepak A, O'Horo JC, Schulz L. Decreasing ICU-associated Clostridioides difficile infection through fluoroquinolone restriction, the FIRST trial: a study protocol. BMJ Open. 2021 Jun 29;11(6):e046480. doi: 10.1136/bmjopen-2020-046480. PMID 34187821